CLINICAL TRIAL: NCT01250951
Title: 1 Year, Open-label Multicenter Evaluation of Efficacy, Safety of Deferasirox in Patients MDS, Thalassemia and Rare Anemia Types Having Transfusion-induced Iron Overload.
Brief Title: This Study Will Evaluate Efficacy and Safety of Deferasirox in Patients With Myelodysplastic Syndromes (MDS), Thalassemia and Rare Anemia Types Having Transfusion-induced Iron Overload.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670ARU01
Record Dates: First submitted 2010-11-11; First posted 2010-12-01 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Myelodysplastic Syndrome; Thalassemia
Keywords: Iron Overload; hemotranfusion; deferasirox; ferritin; Rare anemia; Transfusional Iron Overload
MeSH Terms: conditions — Myelodysplastic Syndromes; Thalassemia; Iron Overload | interventions — Deferasirox

ARMS (1):
- Deferasirox (Experimental)
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox
  Other Names: ICL670

SUMMARY:
This study will evaluate the efficacy and safety of deferasirox in patients with MDS, thalassemia and rare anemia patients with transfusion iron overload.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 2 years
2. Primary Diagnosis: Myelodysplastic Syndrome (presenting with low or intermediate-1 IPSS risk), thalassemia or rare anemias patients (anemia Diamond-Blackfan, Fanconi's anemia, Sideroblastic anemia, Red cell aplasia)
3. ECOG Performance Status ≤ 2
4. Transfusion overload confirmed with ferritin level >1000 µg/l.
5. No severe concomitant uncontrolled disease (uncontrolled diabetes mellitus, heart failure, renal failure).
6. Serum creatine level > ULN
7. No proteinuria
8. Liver enzymes level < 5 ULN.
9. No pregnancy or lactation
10. Signed informed consent by adults. In case inclusion of children under 18 years old, the informed consent should be signed by parents.

Exclusion Criteria:

1. Age < 2 years
2. No iron overload (Ferritin level <1000 µg/l).
3. Primary iron overload (hereditary hemochromatosis)
4. Severe concomitant disease (uncontrolled diabetes mellitus, heart failure, renal failure)
5. Elevated serum creatinine > ULN or/and proteinuria
6. Liver enzymes level >5 ULN.
7. Pregnancy or lactation.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
changes in ferritin level, compared to baseline, in patients with transfusion-induced iron overload treated with Exjade | Baseline assessment is followed by monthly assessments for up to 1 year

SECONDARY OUTCOMES:
changes in clinical manifestations of iron overload by means of echocardiogram (ECHO), electrocardiogram (ECG), routine laboratory assessments and physical examination | Baseline assessment is followed by monthly assessments for up to 1 year.
changes in iron overload evidence on cardiac and liver magnetic resonance imaging (MRI) T2*, compared to baseline, in patients with transfusion-induced iron overload treated with Exjade | at baseline and 1 at year (at the end of study).
Number of participants with adverse events. Safety is evaluated through the continuous monitoring and recording of adverse events, as well as though routine laboratory assessments and physical examination. | From the start of study up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg

REFERENCES:
- [Result] Pennell DJ, Porter JB, Cappellini MD, El-Beshlawy A, Chan LL, Aydinok Y, Elalfy MS, Sutcharitchan P, Li CK, Ibrahim H, Viprakasit V, Kattamis A, Smith G, Habr D, Domokos G, Roubert B, Taher A. Efficacy of deferasirox in reducing and preventing cardiac iron overload in beta-thalassemia. Blood. 2010 Mar 25;115(12):2364-71. Epub 2009 Dec 8. Cappellini MD, Porter J, El-Beshlawy A, Li CK, Seymour JF, Elalfy M, Gattermann N, Giraudier S, Lee JW, Chan LL, Lin KH, Rose C, Taher A, Thein SL, Viprakasit V, Habr D, Domokos G, Roubert B, Kattamis A; EPIC Study Investigators. Tailoring iron chelation by iron intake and serum ferritin: the prospective EPIC study of deferasirox in 1744 patients with transfusion-dependent anemias. Haematologica. 2010 Apr;95(4):557-66. Epub 2009 Nov 30.
- See also: Deferasirox — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a606002.html
- See also: Thalassemia — http://www.nlm.nih.gov/medlineplus/thalassemia.html
- See also: Myelodisplastic Syndrome — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3aproject=medlineplus&v%3asources=medlineplus-bundle&query=myelodysplastic%20syndrome&
- See also: Related Info — http://www.medlit.ru/journal/annotation/1375